CLINICAL TRIAL: NCT02779127
Title: Impact of Ban on Smoking in Pubs, Restaurants and Nightclubs on Endothelial Function in Workers : Evaluation of Endothelial Vasomotoricity Before and After Cessation of Exposure to Passive Smoking : DILATER Study
Brief Title: Impact of Ban on Smoking in Pubs, Restaurants and Nightclubs on Endothelial Function in Workers
Acronym: DILATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 07 269 03
Record Dates: First submitted 2016-03-09; First posted 2016-05-20 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Smoking
Keywords: Smoking; Endothelium; Passive smoking
MeSH Terms: conditions — Smoking | interventions — Independent Medical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): Subjects exposed to passive smoking at least 1 hour per day since 1 year, non active smokers, non exposed to passive smoking at home
  Subject will receive a complete medical follow-up including : medical examination, medical interrogatory, general bioassay, specific bioassay and endothelial function evaluation
  Interventions: Other: Medical interrogatory; Other: Medical examination; Other: Specific bioassay; Other: Endothelial function evaluation; Other: General bioassay
- Control (Other): Subjects non expose to passive smoking at home or at work, non active smokers
  Subject will receive a complete medical follow-up including : medical examination, medical interrogatory, general bioassay, specific bioassay and endothelial function evaluation
  Interventions: Other: Medical interrogatory; Other: Medical examination; Other: Specific bioassay; Other: Endothelial function evaluation; Other: General bioassay

INTERVENTIONS:
Other: Medical interrogatory — Cardiovascular risk, medical history, known pathologies and actual treatments are evaluated
Other: Medical examination — Systolic blood pressure, diastolic blood pressure, cardiac frequency, pulse palpation, hearth and pulmonary auscultation
Other: Specific bioassay — Exhaled carbon monoxide measure and nicotine in the urine are evaluated
Other: Endothelial function evaluation — Endothelial function evaluation done by echotracking determining the basale flow mediated dilatation
Other: General bioassay — Fasting bioassay evaluating total cholesterol, low density lipoproteins, high density lipoproteins, triglycerides, creatine, transaminases, gamma glutamyl transferases, fibrinogen, reactive protein C, blood count and sedimentation rate.

SUMMARY:
Endothelium is considered a real member, so it is contributing to determine the vascular homeostasis. The presence of endothelial dysfunction, evaluated in peripheral arteries by non-invasive study of the variation of gauge of the brachial artery as a result of post-ischemic hyperemia (FMD), is predictive of occurrence of major cardiovascular events. Several recent studies have shown that passive smoking is correlated with endothelial dysfunction and, therefore, non-smokers exposed subjects to passive smoking, have an increased risk of occurrence cardiovascular pathologies. From January 2008, a ministerial decree will ban smoking in bars, restaurants and nightclubs. The impact of exposure end to smoking in non-smoking subjects, as part of a prospective study and controlled, has never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject exposed at least one hour per day to passive smoking at work during at 1 year minimum for intervention arm and non exposed to passive smoking for control group.
* Subject having signed informed consent
* Subject with social security insurance or equivalent

Exclusion Criteria:

* Exposition to passive smoking at home
* Active smokers (at least 1 cigarette per day or having drawn up active smoking for less than a month)
* Medical history of homozygote familial hypercholesterolemia
* Usage of lipid lowering treatment in the month before the inclusion
* Hepatic active pathology or hepatocellular insufficiency
* Severe kidney disease (with creatine clearance less than 30 ml per minute)
* Evolutive cancer
* Usage of concomitant treatment as : insulin, nitro-derivatives and statins
* Medical history of alcoholism or drug use last year
* Medical history of permanent systolic hypotension (systolic blood pressure less than 90 mmHg) or non controled hypertension (systolic blood pressure higher than 200 mmHg and diastolic blood pressure 110 mmHg)
* Active cardiovascular disease
* Psychological or medical conditions incompatible with the study according to investigator opinion
* Participation to another study with experimental product or subject having received an study treatment within 4 weeks before inclusion
* Impossibility to follow the study procedure
* Pregnancy and breastfeeding
* Subject protected by french law

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Comparison of Endothelial function between two groups of non smoking workers exposed or not to passive smoking at work before and after interdiction of smoking decree as assessed by mean change in dilatation percentage of brachial artery. | change between Day 0 and Day 90
  Percentage of dilation of the brachial artery after test ischemia will be compared at the start and at the end of the study (Day 90)

SECONDARY OUTCOMES:
Determination of flow mediated dilatation in non smokers patient as assessed by mean change in dilatation percentage of brachial artery. | change between Day 0 and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra BURA-RIVIERE, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No